CLINICAL TRIAL: NCT04178655
Title: Range of Motion and Function Following Primary Repair of Traumatic Zone 1 or Zone 2 Digit Flexor Tendon Injuries - Impact of Tranexamic Acid Use - A Prospective Study
Brief Title: Tranexamic Acid Effect on Digit Function Following Primary Repair of Traumatic Digit Flexor Tendon Injuries
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Sorin Daniel Iordache, Hand Surgery Unit Director, Rabin Medical Center, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0219-19-RMC
Record Dates: First submitted 2019-11-01; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Tendon Injury - Hand
Keywords: Tendon Injury, Tranexamic Acid
MeSH Terms: conditions — Tendon Injuries | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic Acid Treatment (Experimental): 1 GRAM TRANEXAMIC ACID INTRAVENOUS BOLUS ONCE PRIOR TO SKIN INCISION AND TOURNIQUET INFLATION
  Interventions: Drug: Tranexamic acid injection
- Placebo (Placebo Comparator): 10 MILILITERS 0.9% NORMAL SALINE INTRAVENOUS BOLUS ONCE PRIOR TO SKIN INCISION AND TOURNIQUET INFLATION
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: Tranexamic acid injection — 1 GRAM TRANEXAMIC ACID INTRAVENOUS BOLUS ONCE PRIOR TO SKIN INCISION AND TOURNIQUET INFLATION
  Arms: Tranexamic Acid Treatment
Drug: PLACEBO — 10 MILILITERS 0.9% NORMAL SALINE INTRAVENOUS BOLUS ONCE PRIOR TO SKIN INCISION AND TOURNIQUET INFLATION
  Arms: Placebo

SUMMARY:
This study evaluates the effect of pre-operative treatment with IV Tranexamic Acid on post-operative digit function, in patients that underwent surgical repair of traumatic zone 1 or zone 2 digit flexor tendon tear.

DETAILED DESCRIPTION:
Peritendinous adhesions following repair of digital flexor tendons are a major postoperative complication, due to loss of motion and the functional disability that they cause.

Patients who will present to Rabin Medical Center with acute traumatic Zone 1 or Zone 2 Digit flexor tendon injury, will be recruited to the study, given the patients' informed consent.

Patients recruited to the study will be randomly assigned to either the study group or control group:

1. Study Group - Intra-venous Tranexamic acid treatment
2. Control Group - Placebo (Intra-venous normal saline 0.9%)

All patients will be treated operatively with primary repair of the lacerated flexor tendon.

All patients will be treated post-operatively with early controlled mobilization according to the Duran Protocol.

Randomization of the patients will take place before surgery, in the following manner:

half of the study population will be treated with IV Tranexamic Acid , the other half will be treated with or IV Normal Saline as Placebo.

Either Tranexamic Acid or IV Normal Saline will be administered by the anesthesiologist present in the operating room, prior to tourniquet inflation.

Each patient will be assigned a serial number, and 2 envelopes allocated to that serial number will be prepared in advance. The first envelope will be attached to the patient's file, and be given only to the anesthesiologist in the operating room. The second envelope assigned to the patient will remain closed until the end of the study, along with the study's documents.

All study patients and hand surgeons will be blinded to the treatment received by the study population.

Post-Operative measurements will be made by an orthopedic surgeon or occupational therapist, which will also be blinded to the treatment received by the study population.

To ensure confidentiality, all study documents and data will be kept inside a locked closet, in a locked room in the orthopedic department

ELIGIBILITY:
Inclusion Criteria:

* Patients that will undergo surgical repair of traumatic zone 1 or zone 2 digit flexor tendon tears

Exclusion Criteria:

* Age < 18
* Pregnant Women
* Patients that presented 3 weeks or later after the injury
* Medical history positive for Rheumatic disease
* Current active treatment with anti-coagulation medications
* Injury to more than one finger
* Presence of a fracture in the affected finger
* Presence of a nerve injury in the affected finger that won't enable early use and activation in early rehabilitation protocol
* Mangled extremity injury, degloving injury or other soft tissue injuries that won't enable primary closure of skin
* Previous tear of the affected tendon
* Degenerative tear of flexor tendon
* Tendon tear secondary to infection
* Previous injuries to contralateral side causing dysfunction and/or decreased fingers' range of motion
* Contraindications to Tranexamic acid treatment:

  * Known hypersensitivity to tranexamic acid or to any other ingredient of the preparation.
  * Patients with thromboembolic disease.
  * Patients with active intravascular clotting.
  * Severe renal failure because of risk of accumulation.
  * Patients with subarachnoid hemorrhage
  * Patients with acquired defective color vision

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Anatomic Result at 4-Months post-operatively | Documentation will take place pre-operatively, and 4-months post-operatively during out-patient clinic follow-up.
  Measurement of the anatomical outcome for both Zone1 and Zone 2 tears will be achieved by measuring the Total Active Motion (TAM) using the American Society for Surgery of the Hand Criteria (ASSH).
  Active flexion of the MCPJ, PIP and DIP joints are measured in degrees, and summed. Extension deficits in these joints are measured in degrees, summed, and deducted from the flexion measurements. The full TAM of a finger is 260 degrees: MCPJ 85 degrees, PIPJ 110 degrees and DIPJ 65 degrees The TAM of the affected side can be compared to the normal contralateral side, and expressed as percentage of return of motion.
  The Change of the TAM from baseline will be recorded for at the planned serial follow-ups, as described below.

SECONDARY OUTCOMES:
Anatomic Result at 2-weeks and 8-weeks post-operatively | Serial documentation will take place pre-operatively, and post-operatively during out-patient clinic follow-ups on a planned basis at 2-weeks and 8-weeks post-operatively.
  Measurement of the anatomical outcome for both Zone1 and Zone 2 tears will be achieved by measuring the Total Active Motion (TAM) using the American Society for Surgery of the Hand Criteria (ASSH).
  Active flexion of the MCPJ, PIP and DIP joints are measured in degrees, and summed. Extension deficits in these joints are measured in degrees, summed, and deducted from the flexion measurements. The full TAM of a finger is 260 degrees: MCPJ 85 degrees, PIPJ 110 degrees and DIPJ 65 degrees The TAM of the affected side can be compared to the normal contralateral side, and expressed as percentage of return of motion.
  The Change of the TAM from baseline to each post-operative follow up will be recorded.
Extent of finger and hand swelling | Serial documentation will take place pre-operatively, and post-operatively during out-patient clinic follow-ups on a planned basis: 2-weeks, 8-weeks, and 4-months post-operatively.
  Estimation of finger and hand swelling will be achieved by calculating a Swelling-Ratio (SR). Direct measurement of the circumference of both the affected and unaffected finger and hand palm will be made. Finger circumference will be measured in two anatomic locations: the middle of both the proximal and middle phalanx. Hand circumference will be measured on the level of the distal palmar crease. Above measurements will be documented in centimeters.
  The SR will be calculated by dividing the circumference of the affected side by the circumference of the unaffected side.
Strength Result | Serial documentation will take place post-operatively during out-patient clinic follow-ups on a planned basis: 2-weeks, 8-weeks, and 4-months post-operatively.
  Grip Strength is a widely-used clinical assessment tool , which gives a good global assessment of muscle strength, and delineates the impact of tendon injury on overall strength.
  After flexor tendon repair, impairments are more common in isolated finger flexion than in overall handgrip strength. overall grip strength is the mainstay of strength assessment.
  There are several standardized protocols to assess grip strength, one is performing the measurement with the elbow flexed 90 degrees, the forearm in neutral, and the Patient gripping the Jamar dynamometer at the second handle position. Estimation of hand grip strength will be achieved by calculating a Grip Strength-Ratio (GSR). Direct measurement of the Grip strength of both the affected and unaffected hands will be made. Above measurements will be documented in kilograms.
  The GSR will be calculated by dividing the grip strength of the affected hand by the grip strength of the unaffected side.
Functional Result - DASH Score | Serial documentation will take place post-operatively during out-patient clinic follow-ups on a planned basis: 2-weeks, 8-weeks, and 4-months post-operatively.
  Functional Evaluation will be achieved using the DASH (Disabilities of the Arm, Shoulder and Hand) Questionnaire.
  The DASH Score is the current most practiced scale for upper extremity functionality, and was extensively validated in numerous studies.
  The Scale ranges from 0 (no disability) to 100 (most severe disability).
Functional Result - PRWE Score | Serial documentation will take place post-operatively during out-patient clinic follow-ups on a planned basis: 2-weeks, 8-weeks, and 4-months post-operatively.
  Functional Evaluation will be achieved using the PRWE (Patient-Rated Wrist Evaluation) Questionnaire.
  The PRWE was originally developed in 1998 as a measure of patient-rated pain and disability, following Distal Radius or Scaphoid Fractures.
  The Scale ranges from 0 (no disability) to 100 (most severe disability).

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: within 6 months of study completion
Access Criteria: requests will be reviewed by an external independent review panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Pulos N, Bozentka DJ. Management of complications of flexor tendon injuries. Hand Clin. 2015 May;31(2):293-9. doi: 10.1016/j.hcl.2014.12.004. Epub 2015 Feb 28. PMID 25934203
- [Background] Legrand A, Kaufman Y, Long C, Fox PM. Molecular Biology of Flexor Tendon Healing in Relation to Reduction of Tendon Adhesions. J Hand Surg Am. 2017 Sep;42(9):722-726. doi: 10.1016/j.jhsa.2017.06.013. Epub 2017 Jul 12. PMID 28709791
- [Background] Khanna A, Friel M, Gougoulias N, Longo UG, Maffulli N. Prevention of adhesions in surgery of the flexor tendons of the hand: what is the evidence? Br Med Bull. 2009;90:85-109. doi: 10.1093/bmb/ldp013. Epub 2009 Apr 24. PMID 19395470
- [Background] Sharma P, Maffulli N. Tendon injury and tendinopathy: healing and repair. J Bone Joint Surg Am. 2005 Jan;87(1):187-202. doi: 10.2106/JBJS.D.01850. PMID 15634833
- [Background] Ishiyama N, Moro T, Ohe T, Miura T, Ishihara K, Konno T, Ohyama T, Kimura M, Kyomoto M, Saito T, Nakamura K, Kawaguchi H. Reduction of Peritendinous adhesions by hydrogel containing biocompatible phospholipid polymer MPC for tendon repair. J Bone Joint Surg Am. 2011 Jan 19;93(2):142-9. doi: 10.2106/JBJS.I.01634. PMID 21248211
- [Background] Murphy PG, Loitz BJ, Frank CB, Hart DA. Influence of exogenous growth factors on the synthesis and secretion of collagen types I and III by explants of normal and healing rabbit ligaments. Biochem Cell Biol. 1994 Sep-Oct;72(9-10):403-9. doi: 10.1139/o94-054. PMID 7605612
- [Background] Lin ZX, Woolf SK. Safety, Efficacy, and Cost-effectiveness of Tranexamic Acid in Orthopedic Surgery. Orthopedics. 2016 Mar-Apr;39(2):119-30. doi: 10.3928/01477447-20160301-05. Epub 2016 Mar 4. PMID 26942474
- [Background] Aguilera X, Martinez-Zapata MJ, Hinarejos P, Jordan M, Leal J, Gonzalez JC, Monllau JC, Celaya F, Rodriguez-Arias A, Fernandez JA, Pelfort X, Puig-Verdie Ll. Topical and intravenous tranexamic acid reduce blood loss compared to routine hemostasis in total knee arthroplasty: a multicenter, randomized, controlled trial. Arch Orthop Trauma Surg. 2015 Jul;135(7):1017-25. doi: 10.1007/s00402-015-2232-8. Epub 2015 May 7. PMID 25944156
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Gandhi R, Evans HM, Mahomed SR, Mahomed NN. Tranexamic acid and the reduction of blood loss in total knee and hip arthroplasty: a meta-analysis. BMC Res Notes. 2013 May 7;6:184. doi: 10.1186/1756-0500-6-184. PMID 23651507
- [Background] McConnell JS, Shewale S, Munro NA, Shah K, Deakin AH, Kinninmonth AW. Reduction of blood loss in primary hip arthroplasty with tranexamic acid or fibrin spray. Acta Orthop. 2011 Dec;82(6):660-3. doi: 10.3109/17453674.2011.623568. Epub 2011 Oct 17. PMID 21999623
- [Background] Niskanen RO, Korkala OL. Tranexamic acid reduces blood loss in cemented hip arthroplasty: a randomized, double-blind study of 39 patients with osteoarthritis. Acta Orthop. 2005 Dec;76(6):829-32. doi: 10.1080/17453670510045444. PMID 16470437
- [Background] Oremus K, Sostaric S, Trkulja V, Haspl M. Influence of tranexamic acid on postoperative autologous blood retransfusion in primary total hip and knee arthroplasty: a randomized controlled trial. Transfusion. 2014 Jan;54(1):31-41. doi: 10.1111/trf.12224. Epub 2013 Apr 25. PMID 23614539
- [Background] Frueh FS, Kunz VS, Gravestock IJ, Held L, Haefeli M, Giovanoli P, Calcagni M. Primary flexor tendon repair in zones 1 and 2: early passive mobilization versus controlled active motion. J Hand Surg Am. 2014 Jul;39(7):1344-50. doi: 10.1016/j.jhsa.2014.03.025. Epub 2014 May 5. PMID 24799144
- [Background] Jansen CW, Watson MG. Measurement of range of motion of the finger after flexor tendon repair in zone II of the hand. J Hand Surg Am. 1993 May;18(3):411-7. doi: 10.1016/0363-5023(93)90083-f. PMID 8515007
- [Background] Strickland JW, Glogovac SV. Digital function following flexor tendon repair in Zone II: A comparison of immobilization and controlled passive motion techniques. J Hand Surg Am. 1980 Nov;5(6):537-43. doi: 10.1016/s0363-5023(80)80101-8. PMID 7430595
- [Background] Tang JB. Outcomes and evaluation of flexor tendon repair. Hand Clin. 2013 May;29(2):251-9. doi: 10.1016/j.hcl.2013.02.007. PMID 23660061
- [Background] Elliot D, Harris SB. The assessment of flexor tendon function after primary tendon repair. Hand Clin. 2003 Aug;19(3):495-503. doi: 10.1016/s0749-0712(03)00028-3. PMID 12945647
- [Background] MacDermid JC. Measurement of health outcomes following tendon and nerve repair. J Hand Ther. 2005 Apr-Jun;18(2):297-312. doi: 10.1197/j.jht.2005.02.009. PMID 15891987
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] Hoang-Kim A, Pegreffi F, Moroni A, Ladd A. Measuring wrist and hand function: common scales and checklists. Injury. 2011 Mar;42(3):253-8. doi: 10.1016/j.injury.2010.11.050. Epub 2010 Dec 15. PMID 21159335
- [Background] Libberecht K, Lafaire C, Van Hee R. Evaluation and functional assessment of flexor tendon repair in the hand. Acta Chir Belg. 2006 Sep-Oct;106(5):560-5. doi: 10.1080/00015458.2006.11679952. PMID 17168270
- [Background] Dacombe PJ, Amirfeyz R, Davis T. Patient-Reported Outcome Measures for Hand and Wrist Trauma: Is There Sufficient Evidence of Reliability, Validity, and Responsiveness? Hand (N Y). 2016 Mar;11(1):11-21. doi: 10.1177/1558944715614855. Epub 2016 Jan 13. PMID 27418884
- [Background] MacDermid JC, Turgeon T, Richards RS, Beadle M, Roth JH. Patient rating of wrist pain and disability: a reliable and valid measurement tool. J Orthop Trauma. 1998 Nov-Dec;12(8):577-86. doi: 10.1097/00005131-199811000-00009. PMID 9840793